CLINICAL TRIAL: NCT00213590
Title: A Multicentric, Randomized, Opened Study to Evaluate Efficacy on Renal Function of an Immunosuppressant Regimen Based on Cyclosporine A Dose Reduction in Combination With Mycophenolate Mofetil, From the Second Year of Renal Transplantation
Brief Title: Renal Function Evaluation After Reduction of Cyclosporine A Dose in Renal Transplant Patients
Acronym: DICAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1998/081/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Kidney Transplantation; Primary Prevention; Kidney Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): the usual-exposure group, the cyclosporine AUC0-12h target was 4.3 (3.5 to 4.8, range) mg•h/L
- 2 (Experimental): the low-exposure group the cyclosporine AUC0-12h target was 50% usual target or 2.2 (2.0 to 2.6, range) mg•h/L
  Interventions: Drug: cyclosporine A

INTERVENTIONS:
Drug: cyclosporine A — The usual-exposure level was based on the mean area-under-the-concentration-time curve (AUC0-12h). In the usual-exposure group, the cyclosporine AUC0-12h target was 4.3 (3.5 to 4.8, range) mg•h/L and in the low-exposure group the target was 50% or 2.2 (2.0 to 2.6, range) mg•h/L. Ranges were asymmetrical for safety reasons, i.e., to prevent the occurrence of rejection in the low-exposure arm and nephrotoxicity in the usual-exposure arm.The AUC 0-12h was estimated using a Bayesian estimator and a three-point limited sampling strategy (0, 1, and 3 hours). A computer program was used to calculate the dose adjustment required to reach the therapeutic target. Doses were adjusted in increments of 25% to reach the target within 2 months. Cyclosporine AUC0-12h was determined every 2 months.
  Other Names: cyclosporine microemulsion Neoral Novartis Basel Switzerland
  Arms: 2

SUMMARY:
The purpose of the study is to show the efficacy of reduction of cyclosporine A exposure measured by the area under the curve by Bayesian estimator on the primary prevention of degradation of the renal function in renal transplant recipients

DETAILED DESCRIPTION:
Study population Eligible patients were 18 to 75 years of age and primary or secondary renal transplant recipients in their second year posttransplant with stable serum creatinine levels (i.e., < 20% variation for the previous 3 months). All patients must have received induction therapy, been corticosteroid-free for at least 3 months, and receiving combination maintenance therapy consisting of cyclosporine (trough level, 125 to 175 ng/mL) and mycophenolate mofetil (CellCept, F. Hoffmann- La Roche AG, Basel, Switzerland) 2 g daily.

Patients at either low or high risk of graft dysfunction were ineligible; a majority of the participating centers maintained low immunological risk patients on cyclosporine alone and those with a high risk of graft dysfunction were usually maintained on corticosteroids. For this study, low risk was defined as the presence of the following: zero or one acute rejection episode with a return of renal function to previous levels after corticosteroid treatment, panel-reactive antibody titer <25%, serum creatinine level <125 µmol/L, age >25 years, and donor age <40 years. High risk was defined as the presence of at least one of the following: a serum creatinine level >250 µmol/L, proteinuria >1 g/day, panel-reactive antibody titer >80%, >1 episode of T-cell-mediated rejection or at least one episode of antibody-mediated rejection posttransplant, or the presence of vasculitis or systemic lupus erythematosus which usually were treated with corticosteroids.

Other exclusion criteria were evidence of systemic infection or malignancy within the previous 5 years (except adequately treated nonmetastatic basal or squamous cell carcinoma of the skin), leukocyte count <2.5x103/µL, hemoglobin <80 g/dL, platelet count <100x103/µL, severe intestinal disorders, pregnancy, breast feeding, current immunosuppressive treatment with drugs other than cyclosporine and mycophenolate mofetil. Women of childbearing age were required to use adequate contraception during treatment with mycophenolate mofetil and for six weeks after its discontinuation.

Study Endpoints The primary endpoint was the proportion of patients with treatment failure (failure to prevent kidney dysfunction) at 24 months, which was a composite of graft loss, histologically confirmed acute rejection or cyclosporine toxicity, or a > 15% increase in the mean serum creatinine level from the baseline assessment. The mean of the current and two previous serum creatinine levels was used to determine the level at baseline, the level at the nadir (the time of the lowest serum creatinine measurement),and the level at 2 years.

The secondary endpoints included the change in estimated glomerular filtration rate (eGFR) from baseline calculated using the four-variable equation from the Modification of Diet in Renal Disease (MDRD) Study; blood pressure, urinary protein, and lipid levels; severe adverse events such as infection requiring hospitalization, neoplasia, or lymphoma; and graft and patient survival.

Study Follow-up and Procedures Weight, blood pressure after a 10-minute rest, serum creatinine and glucose levels, a complete blood cell count, and urinary protein levels were measured, and the use of immunosuppressive, antihypertensive, and lipid-lowering drugs was recorded at baseline and every 2 months. Serum lipid levels were measured at baseline and every 6 months. Gynecologic and dermatologic examinations were performed at baseline and yearly. Adverse events were recorded.

Renal biopsies were performed when creatinine levels increased > 20% relative to the nadir or when proteinuria was >1 g/day. The nadir level was used as a reference point to obviate the risk of missing the diagnosis of rejection in the low-exposure arm; serum creatinine levels usually fell after the initiation of a low exposure regimen. Biopsies were classified using Banff 1997 criteria by four senior pathologists blinded to the clinical information. CNI-associated nephrotoxicity was graded mild, moderate, or severe according to the Banff 1997 chronicity rejection scores.

ELIGIBILITY:
Inclusion Criteria:

* first or second renal graft
* cadaveric renal graft
* second year of renal transplantation
* stable renal function
* moderate renal dysfunction risk
* bitherapy with cyclosporine A and mycophenolate mofetil
* corticosteroid withdrawal since 3 months at less

Exclusion Criteria:

* 2 or more acute rejection episodes
* PRA> 80%
* serum creatinine> 250µmol/L
* 24-hour proteinuria > 1g
* humoral rejection
* vasculitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2000-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
renal function at two years | every two months

SECONDARY OUTCOMES:
proteinuria | every two months
hypertension | every two months
hemodialysis | at any time during the study period
nephrotoxicity | at any time during the study period
chronic renal dysfunction | at two years
biopsy proven late acute rejection | at any time during the study period
dyslipidemia | every six months
patient survival | at two years
graft survival | at two years
severe infection with hospitalisation | at any time during the study period
post transplant lymphoproliferative disorder | at any time during the study period
cutaneous carcinoma | every year
area under the concentration-time of cyclosporine A | every two months
area under the concentration-time of mycophenolate mofetil | at month 0 6 12 and 24
biodisponibility of mycophenolate mofetil after reduction of cyclosporine A exposure | at month 6 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle ETIENNE, MD, Principal Investigator — University Hospital, Rouen